CLINICAL TRIAL: NCT06426784
Title: Perfusion Index as a Predictor of Hypotension Following Sub-arachnoid Block Among Patients Undergoing Lower Segment Caesarean Section
Status: Completed | Type: Observational
Sponsor: Muhammad Haroon Anwar (Other Government)
Collaborators: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Sponsor-Investigator, Muhammad Haroon Anwar, Principal Investigator, Department of Anaesthesia and Critical Care Medicine, Pakistan Institute of Medical Sciences
Organization: Pakistan Institute of Medical Sciences (Other Government)
Other Study IDs: F-5-2/2024(ERRB)/PIMS
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Hypotension; Hypotension on Induction; Spinal Anesthetics Causing Adverse Effects in Therapeutic Use
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Low Perfusion index: Pregnant patients having baseline perfusion index less than 3.5 will be enrolled into this group.
- High Perfusion index: Pregnant patients having baseline perfusion index ≥ 3.5 will be enrolled into this group.

SUMMARY:
C-section is one of the commonly performed surgical procedures. During this surgical procedure the surgeon cuts into uterine cavity through abdominal wall and takes out the baby. This is done by by making the lower half body of the patient numb by injecting local anesthesia drugs into the space surrounding the spinal cord. This allows the mother to remain awake and immediately bond with the baby once it gets delivered. Also this technique provides effective pain relief both during and after the surgery. However like any other technique or drug it is associated with a number of side effects. The most important being fall in blood pressure. There are numerous ways to treat it. However if one is able to predict fall in blood pressure before administration of anesthetic technique one can easily prevent it. One of the recently discovered novel way to predict fall in blood pressure is Perfusion index which is calculated by Pulse oximeter. It is a device use to check amount of oxygen in blood and heart rate. Perfusion index refers to the total amount of blood present in the limbs of the person. Once we administer drug in the space surrounding the spinal cord the amount of blood in the limbs increases while the amount returning to heart decreases which ultimately results in less amount of blood being pumped out by heart resulting in fall in blood pressure. Therefore theoretically those individuals who have a high baseline Perfusion index will more likely to develop low blood pressure. This study aims to identify the cut off value of perfusion index to predict fall in blood pressure.

DETAILED DESCRIPTION:
Spinal anesthesia is employed to provide excellent surgical conditions in case of C-Section. It is the anesthetic technique of choice among obstetric patients. However it is associated with sympathectomy which reduces the venous return and ultimately causes hypotension. This hypotension is mainly due to redistribution of blood volume to the peripheral compartment. Perfusion index which is measured by Pulse Oximetery is a ratio of pulsatile to non-pulsatile blood in the peripheral compartment of the body. As spinal anesthesia causes sympathectomy, peripheral blood volume increases. As a result perfusion index value should rise. This will then co-relate with hypotension. In simple terms those individuals who have a high baseline Perfusion index value will more likely to develop hypotension. This study aims to identify the baseline perfusion index value which co-relates with development of hypotension following sub-arachnoid block for C-section.

ELIGIBILITY:
Inclusion Criteria:

* ASA class II and III
* Elective LSCS under sub-arachnoid block
* Age 18-35 years

Exclusion Criteria:

* Hypertensive disorders of pregnancy
* Autonomic neuropathy
* Fetal distress
* NPO >8h
* Lack of maintenance fluid or oral clear fluid intake during NPO period.
* BMI > 35 kg/m2
* Patients requiring Vasopressor and Ionotropic support.

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Pregnant females undergoing elective Lower segment caesarean section
Study Population: Pregnant females undergoing elective lower segment caesarean section under spinal anesthesia at Pakistan Institute of Medical sciences will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-05-27 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of hypotension | Intra-operative peroid
  Number of episodes of hypotension among both groups will be compared.

SECONDARY OUTCOMES:
Baseline perfusion index as a predictor of hypotension | Intra operative peroid
  Sensitivity and specificity of baseline perfusion index to predict intra-operative hypotension following sub-arachnoid block

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Haroon Anwar, MBBS, Principal Investigator — Department of Anesthesia and Critical Care, Pakistan Institute of Medical Sciences, Islamabad
Locations (1):
- Deparment of Anesthesia and Critical Care Medicine, Pakistan Institute of Medical Sciences, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lal J, Bansal T, Bhardwaj S, Jain M, Singh AK. A study to evaluate perfusion index as a predictor of hypotension following spinal anesthesia for caesarean section. J Anaesthesiol Clin Pharmacol. 2022 Apr-Jun;38(2):294-299. doi: 10.4103/joacp.JOACP_385_20. Epub 2022 Jun 16. PMID 36171921